CLINICAL TRIAL: NCT05748431
Title: The Outcome of Percutaneous Balloon Pulmonary Valvuloplasty in Pediatrics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Tarek Mohammed Hafez, Principle investigator, Assiut University
Other Study IDs: 75
Record Dates: First submitted 2022-08-23; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Balloon Pulmonary Valvuloplasty in Pulmonary Valvular Stenosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
evaluation the outcome of percutaneous balloon pulmonary valvuloplasty in children with valvular pulmonary stenosis at the Pediatric Cardiology Unit.

DETAILED DESCRIPTION:
Pulmonary valve stenosis (PS) is a heart valve disorder in which outflow of blood from the right ventricle of the heart is obstructed at the level of the pulmonic valve. Although most commonly diagnosed and treated in the pediatric population, individuals with more severe forms of PS are surviving into adulthood and require ongoing assessment and cardiovascular care. The prevalence of valvular pulmonary stenosis has been reported at 0.6 to 0.8 cases per 1000 live births. When associated with other congenital heart disorder, it occurs in approximately 50% of all born with some kind of congenital heart disease . Pulmonary stenosis can be due to isolated valvular (90%), subvalvular, or peripheral (supravalvular) obstruction, or it may be found in association with congenital heart disorders of some other kind .

Critical pulmonary stenosis (PS) is a life-threatening congenital heart disease which requires immediate treatment . Unlike older children with isolated PS, neonates with critical PS presents with severe cyanosis and the suprasystemic right ventricle (RV) pressure may result in RV dilatation and failure with severe tricuspid regurgitation (TR). Since the discovery of balloon pulmonary valvuloplasty (BPV), it has replaced surgical approach for relieving PS . Femoral vein is the most common venous access for BPV; however, crossing the pulmonary valve using this approach can be difficult, especially in the presence of severe TR and right chambers dilatation . This problem can be overcome by using transjugular approach, yet many operators are reluctant to use this method because of potential complications and lack of data reporting transjugular approach. Balloon pulmonary valvuloplasty (BPV) is a safe and effective treatment for isolated pulmonary valve stenosis . The optimal age or body size for elective BPV depends on an individual's pulmonary valve diameter, transpulmonary pressure gradient, and femoral vessel size. Selecting a balloon with an appropriate profile also affects outcomes. An ideal balloon catheter for BPV in younger, smaller patients would have a low profile with a short, round shoulder to lessen the risk of valvular or vascular injury . Balloon pulmonary valvuloplasty provides long-term relief of stenosis of the pulmonary valve in the majority of patients with moderate to severe pulmonary valve stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Children with valvular pulmonary stenosis confirmed by Echocardiography, and managed with percutaneous balloon pulmonary valvuloplasty

Exclusion Criteria:

* Cases with pulmonary stenosis not candidate for balloon valvuloplasty Cases with pulmonary stenosis associated with other congenital heart diseases

Ages: 1 Day to 6 Years | Sex: All
Age Groups: Child
Study Population: Pediatric Cardiology Unit, Children and Cardiology Assiut University Hospitals
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the outcome of percutaneous ballon pulmonary valvuloplasty in children with pulmonary valvular stenosis at the pediatric cardiology unit | 3 years
  Evaluation depend on Echocariography measurement of pressure gradient pre and post valvuloplasty for about 100 cases of children up to 6 years in the pediatric cardiology y